CLINICAL TRIAL: NCT01398514
Title: Pharmacologic Influence of Escitalopram on the Reduction of Fear Acquisition and Triggered Renewal During Fear Conditioning: a Model for the Prevention and Persistence of Learned Fear and Anxiety in Response to Trauma and Stress
Brief Title: Influence of Escitalopram on Fear Conditioning
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Principal Investigator, Naomi M. Simon, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2008-P-001314
Record Dates: First submitted 2011-07-12; First posted 2011-07-20 (Estimated); Results first posted 2013-09-27 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-06

CONDITIONS: Fear Conditioning
MeSH Terms: interventions — Escitalopram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active medication (Experimental): Escitalopram 10mg/day
  Interventions: Drug: Escitalopram
- Placebo (Placebo Comparator): Matched pill placebo
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram — Escitalopram 10mg/day or matched pill placebo

SUMMARY:
The purpose of the study is to learn how differences in learning under mildly-stressful circumstances may be changed by taking an antidepressant medication. This medication is called Lexapro (Escitalopram). The investigators will also examine the impact of any anxiety, depression, and stress related symptoms on learning processes. The investigators will also look at the response of these symptoms to Lexapro.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female outpatients 18 to 75 years of age
2. Must have no current DSM-IV Axis I diagnosis as measured by the SCID (Structured Clinical Interview for DSM-IV-TR axis 1 disorders) with a trained study investigator. Past history of anxiety disorders, major depressive episodes or substance abuse disorders at least six months prior to baseline are not exclusionary.

Exclusion Criteria:

1. Patients will be excluded from entry into the study for current serious medical conditions or other conditions deemed likely to result in surgery or hospitalization.
2. Patients with a history of trauma resulting in head injury related seizures, or with epilepsy (except a prior history of febrile seizures of infancy which are not exclusionary).
3. Pregnant or lactating women or those of childbearing potential not using medically accepted forms of contraception will be excluded.
4. Concurrent use of other antidepressants, benzodiazepines or antipsychotic medications.
5. Patients with a history of hypersensitivity to escitalopram are excluded.
6. Individuals must have discontinued MAO inhibitors more than 14 days before starting study drug.
7. Additional contraindicated drugs during the study are pimozide, furazolidine, isocarboxazid, lazabemide, and St. John's Wort.
8. Participants meeting DSM-IV or SCID criteria for a substance use disorder in the last six months other than nicotine dependence and those with a positive toxicology screen at baseline consistent with evidence of current substance abuse or dependence as determined by clinical interview.
9. A lifetime history of Bipolar or any psychotic disorder is excluded.
10. Current claustrophobia is exclusionary.
11. Patients currently taking any narcotic will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi M Simon, M.D., M.Sc., Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants free of DSM-IV Axis I disorders with varying levels of subsyndromal anxiety were recruited by advertisements (e.g., postings on Craigslist, postings on Massachusetts General Hospital research participation registry) from March 2009 through April 2011.
Pre-assignment Details: 65 participants signed consent and were screened for enrollment. 10 participants did not meet study entry criteria due to exclusionary psychiatric conditions. Of the 55 eligible participants, 3 withdrew and 1 was lost to follow up. 52 participants were randomly assigned to a treatment arm. Fourteen were excluded from analyses.
Period: Overall Study
Arm/Group | Active Medication | Placebo
Started | 26 | 26
Completed | 18 | 20
Not Completed | 8 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Non-compliance with study procedures | 2 | 0
Not completed — Physiologic non-responsiveness | 1 | 3
Not completed — Failure to show a conditioned response | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Medication | Placebo | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 25 | 26 | 51
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.04 (11.56) | 30.46 (11.46) | 32.25 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 12 | 26
  Male | 12 | 14 | 26
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Physiological Reactivity as Measured by Square-root Transformed Skin Conductance Conditioned Response in Early Extinction Trials 1 to 4
Description: Three-way interaction between group (active vs. placebo), CS (+ vs. -), and trials (1 - 4).
  CS+ refers to the conditioned stimulus associated with the unconditioned stimulus (electric shock). Higher numbers reflect higher skin conductance response to the CS+ (conditioned stimulus).
  CS- refers to the stimulus not associated with the unconditioned stimulus. Higher numbers reflect higher skin conductance response to a CS-.
  Square-root transformed skin conductance conditioned response are reported for trials 1 to 4 of the Early Extinction Phase.
Time Frame: Day 2 of Fear Conditioning Paradigm (15 to 18 days post medication initiation)
Measure: Mean (Standard Error); unit: micro-Siemens (square rooted)
Groups:
- Active Medication CS-: Escitalopram 10mg/day
- Active Medication CS+: Matched pill placebo
Arm/Group | Active Medication CS- | Active Medication CS+ | Placebo CS- | Placebo CS+
Number analyzed (Participants) | 16 | 16 | 18 | 18
micro-Siemens (square rooted)
  Trial 1 | 0.745 (0.130) | 0.853 (0.853) | 0.799 (0.122) | 0.717 (0.123)
  Trial 2 | 0.496 (0.103) | 0.634 (0.114) | 0.386 (0.097) | 0.558 (0.108)
  Trial 3 | 0.544 (0.111) | 0.520 (0.124) | 0.438 (0.105) | 0.787 (0.117)
  Trial 4 | 0.374 (0.110) | 0.361 (0.116) | 0.309 (0.104) | 0.510 (0.109)

2. Primary Outcome: Physiological Reactivity as Measured by Square-root Transformed Skin Conductance Conditioned Response in Acquisition Trials 1 to 5
Description: Three-way interaction between group (active vs. placebo), CS (+ vs. -), and trials (1 - 5).
  CS+ refers to the conditioned stimulus associated with the unconditioned stimulus (electric shock). Higher numbers reflect higher skin conductance response to the CS+ (conditioned stimulus).
  CS- refers to the stimulus not associated with the unconditioned stimulus. Higher numbers reflect higher skin conductance response to a CS-.
  Square-root transformed skin conductance conditioned response are reported for trials 1 to 5 of the Acquisition Phase.
Time Frame: Baseline on Day 1 of Fear Conditioning Paradigm (14 to 17 days post medication initiation)
Measure: Mean (Standard Error); unit: micro-Siemens (square rooted)
Arm/Group | Active Medication CS- | Active Medication CS+ | Placebo CS- | Placebo CS+
Number analyzed (Participants) | 18 | 18 | 20 | 20
micro-Siemens (square rooted)
  Trial 1 | 0.634 (0.093) | 0.574 (0.111) | 0.532 (0.088) | 0.634 (0.105)
  Trial 2 | 0.419 (0.122) | 0.870 (0.113) | 0.428 (0.116) | 0.817 (0.107)
  Trial 3 | 0.230 (0.119) | 0.685 (0.104) | 0.331 (0.112) | 0.856 (0.099)
  Trial 4 | 0.231 (0.086) | 0.626 (0.102) | 0.181 (0.082) | 0.677 (0.096)
  Trial 5 | 0.281 (0.071) | 0.543 (0.118) | 0.144 (0.067) | 0.714 (0.112)

ADVERSE EVENTS:
Time Frame: AEs were assessed in the period following randomization/medication initiation, through the experimental portion of the study (14-17 days post medication initiation), and 7 days following medication discontinuation.
Description: AEs were defined as any untoward or unfavorable medical occurrence in a human subject. SAEs event were defined as any event temporally associated with the subject's participation that: results in death, is life-threatening, results in inpatient hospitalization, results in significant disability, or results in a congenital anomaly or birth defect
Arm/Group | Active Medication | Placebo
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/26
Other Adverse Events (participants affected / at risk) | 13/25 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Medication (N=25) | Placebo (N=26)
Appetite decrease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Tremor / Shakiness (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety / Nervousness (Psychiatric disorders) | 2 (2) | 0 (0)
Jitteriness / Restlessness (Nervous system disorders) | 1 (1) | 2 (2)
Vivid or Disturbing Dreams (General disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 1 (1)
Sedation / Drowsiness (General disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Difficulty Concentrating (Psychiatric disorders) | 1 (1) | 0 (0)
Sexual Dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Insomnia (General disorders) | 3 (3) | 0 (0)
Sweating / Hot Flashes (General disorders) | 1 (1) | 0 (0)
Lightheadedness (Nervous system disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Weightloss (Gastrointestinal disorders) | 1 (1) | 0 (0)
Muscle cramping / spasm (Nervous system disorders) | 0 (0) | 1 (1)
Head cold (General disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor shall require the PI to furnish the sponsor with a copy of any proposed publication at least 60 days prior to submission. The sponsor shall be entitled to review such proposed publications. The PI shall give due regard to the sponsor's comments on the proposed publication. If the sponsor reasonably believes a patent application claiming an invention should be filed prior to such publication, such submission shall not be submitted until applicable patent applications have been filed.